CLINICAL TRIAL: NCT00624130
Title: Open, Randomized, Parallel Multi-center Comparison of Cycle Control and Safety of the Oral Contraceptive Yasmin 20 in a 24-day Regimen vs. Mercilon for 7 Cycles in 440 Healthy Female Volunteers
Brief Title: Yasmin 20 Cycle Control - Yasmin 20 Versus Mercilon in Healthy Female Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91352; 308020
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Contraception
Keywords: Contraception,; Cycle control,; Bleeding pattern
MeSH Terms: interventions — ethinyl estradiol-desogestrel combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Yasmin 20
- Arm 2 (Active Comparator)
  Interventions: Drug: Mercilon

INTERVENTIONS:
Drug: Yasmin 20 — Yasmin 20, 24-d regimen vs Mercilon, Tablet p.o. (oral)
  Arms: Arm 1
Drug: Mercilon — Mercilon, 24-d regimen vs Yasmin 20 , Tablet p.o. (oral)
  Arms: Arm 2

SUMMARY:
The purpose of this study is to compare bleeding pattern of contraceptive Yasmin 20 to a marketed comparator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteer aged 18-35,
* Smokers 18-30

Exclusion Criteria:

* Contraindications for using hormonal contraceptives

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 453 (Actual)
Dates: Start 2004-03; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Cycle control and bleeding pattern | 7 cycles

SECONDARY OUTCOMES:
Pearl index | 7 cycles
Laboratory tests | Screening
Adverse Events | 7 cycles
General Physical and gynecological examinations | Screening
Vital signs | Screening, admission
Body weight | Screening, admission

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Austria (6):
  - Horn
  - Leibnitz, Styria
  - Mödling
  - Sankt Pölten
  - Vienna
  - Wörgl
- Estonia (3):
  - Pärnu
  - Talinn
  - Tartu
- Finland (3):
  - Helsinki
  - Tampere
  - Turku
- Lithuania (2):
  - Kaunas
  - Vilnius

REFERENCES:
- [Result] Anttila L, Neunteufel W, Petraglia F, Marr J, Kunz M. Cycle control and bleeding pattern of a 24/4 regimen of drospirenone 3 mg/ethinylestradiol 20 mug compared with a 21/7 regimen of desogestrel 150 mug/ethinylestradiol 20 mug: a pooled analysis. Clin Drug Investig. 2011;31(8):519-525. doi: 10.2165/11590260-000000000-00000. PMID 21721590
- [Result] Anttila L, Bachmann G, Hernadi L, Kunz M, Marr J, Klipping C. Contraceptive efficacy of a combined oral contraceptive containing ethinyloestradiol 20 mug/drospirenone 3mg administered in a 24/4 regimen: a pooled analysis of four open-label studies. Eur J Obstet Gynecol Reprod Biol. 2011 Apr;155(2):180-2. doi: 10.1016/j.ejogrb.2010.12.037. Epub 2011 Feb 1. PMID 21277674